CLINICAL TRIAL: NCT06491966
Title: Comparative Analysis of Clinical Outcomes and Inflammatory Responses in Viral Versus Bacterial Sepsis: A Retrospective Cohort Study in ICU Patients
Brief Title: Clinical Outcomes and Inflammatory Responses in Viral vs. Bacterial Sepsis
Status: Recruiting | Type: Observational
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Lin Chen, chief physician, Sichuan Provincial People's Hospital
Other Study IDs: SichuanPPHLC03
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Sepsis; Sepsis Bacterial; Viral Sepsis; Inflammatory Response; Cytokine Storm; COVID-19; MODS
MeSH Terms: conditions — Sepsis; Viremia; Cytokine Release Syndrome; COVID-19; Multiple Organ Failure | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- viral sepsis group: The viral sepsis group comprises patients with sepsis secondary to viral infections, specifically COVID-19. Patients in this group were admitted to the ICU of Sichuan Provincial People's Hospital between July 2021 and December 2023 and diagnosed with viral sepsis based on positive RT-PCR results for SARS-CoV-2.
  Interventions: Other: observation
- bacterial sepsis group: The bacterial sepsis group includes patients with sepsis resulting from bacterial infections. These patients were admitted to the ICU of Sichuan Provincial People's Hospital during the same period and diagnosed with bacterial sepsis based on positive bacterial cultures.
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — data collected includes demographic information, clinical outcomes (mortality rate, ICU stay length), inflammatory markers (e.g., IL-2, IL-10, TNF-α), and treatment details (mechanical ventilation, CRRT, ECMO, antibiotics). Culture results, NGS findings, and imaging reports were also documented.

SUMMARY:
This observational cohort study aims to compare clinical outcomes and inflammatory responses between patients with viral sepsis, specifically COVID-19-associated sepsis, and those with bacterial sepsis. Conducted at Sichuan Provincial People's Hospital, the study will retrospectively analyze data from ICU patients admitted between July 2021 and December 2023. The primary objective is to identify reliable biomarkers and diagnostic methods to improve patient outcomes through personalized diagnostic and therapeutic strategies.

DETAILED DESCRIPTION:
Sepsis, a major cause of morbidity and mortality in ICU patients, has garnered increased attention during the COVID-19 pandemic due to the high mortality rates associated with viral sepsis. This study seeks to elucidate the differences in clinical outcomes, inflammatory responses, and treatment strategies between bacterial and viral sepsis. By leveraging a comprehensive dataset of ICU patients diagnosed with sepsis at Sichuan Provincial People's Hospital, the study will retrospectively compare the two sepsis types.

A total of 267 patients diagnosed according to Sepsis 3.0 criteria, including 105 with bacterial sepsis and 162 with viral sepsis (COVID-19 confirmed via RT-PCR), will be included. Key clinical parameters such as mortality rate, length of ICU stay, SOFA scores, and the need for life support measures (mechanical ventilation, CRRT, ECMO) will be analyzed. Additionally, the study will examine cytokine profiles and other inflammatory markers to identify significant differences between the two groups.

The study will utilize advanced statistical methods, including Kaplan-Meier survival analysis, multinomial logistic regression, and ROC curve analysis, to evaluate the predictive power of various biomarkers. The findings are expected to highlight critical factors contributing to the higher mortality observed in viral sepsis and inform the development of targeted treatment strategies. The ultimate goal is to improve diagnostic accuracy and patient outcomes through personalized approaches tailored to the type of sepsis.

Key objectives include understanding the distinct inflammatory responses in bacterial and viral sepsis and identifying reliable biomarkers for differentiation. The study will also evaluate the impact of different treatment regimens, particularly antibiotic use, on clinical outcomes. Insights gained from this research will contribute to the broader understanding of sepsis management and guide future clinical practice and research.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with sepsis according to Sepsis 3.0 criteria.
2. Patients with confirmed bacterial sepsis based on positive bacterial cultures.
3. Patients with confirmed viral sepsis, specifically COVID-19, diagnosed via RT-PCR for SARS-CoV-2 for viral group and negative for bacterial group.
4. Patients aged 18 years and older.
5. Patients admitted to the ICU during the study period.

Exclusion Criteria:

1. Patients with mixed bacterial and viral infections.
2. Patients with sepsis not meeting the Sepsis 3.0 criteria.
3. Patients who received immunomodulatory therapies other than standard treatments (e.g., investigational drugs).
4. Pregnant or breastfeeding women.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU of Sichuan Provincial People's Hospital from July 2021 to December 2023 diagnosed with sepsis according to Sepsis 3.0 criteria.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-07-07 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | 28 days
  The primary outcome measure is the mortality rate of patients diagnosed with sepsis. This measure will compare the 28-day survival rate in the ICU between patients with bacterial sepsis and those with viral sepsis, specifically COVID-19-associated sepsis.
Length of ICU stay | From ICU admission until discharge or death, assessed up to 28 days
  This outcome measure will assess the length of ICU stay for patients diagnosed with sepsis. The comparison will be made between bacterial sepsis and viral sepsis patients, considering the duration of ICU admission from the time of diagnosis until discharge or death.

SECONDARY OUTCOMES:
Levels of key inflammatory markers | baseline (Measured at the time of ICU admission)
  This outcome measure will assess the levels of key inflammatory markers, including IL-2, IL-6, IL-8, IL-10, TNF-α, MYD88, mCD64, and nCD64. The comparison will be made between bacterial and viral sepsis patients to identify significant differences in cytokine profiles and their impact on sepsis outcomes.
Incidence of secondary infections | Assessed from the time of ICU admission up to 28 days or until discharge or death, whichever came first
  This outcome measure will evaluate the incidence of secondary infections in patients diagnosed with sepsis. The focus will be on identifying the occurrence of secondary bacterial or fungal infections in both bacterial and viral sepsis groups, as well as the impact of these infections on patient outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Chen, doctor, Principal Investigator — Sichuan Provincial People's Hospita
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided
At this stage, the decision on whether to make individual participant data (IPD) available to other researchers has not been finalized. Considerations include ethical and privacy concerns, institutional policies, and the potential benefit to the scientific community. If data sharing is implemented in the future, it will comply with relevant regulations and guidelines, ensuring the privacy and confidentiality of the participants. Researchers interested in accessing the IPD may contact the principal investigator for further information and potential collaboration opportunities.

REFERENCES:
- [Derived] Xiong L, Tang H, Xie Q, Fang H, Jing D, Chen L. Immune Signatures Distinguish Pure and Mixed Sepsis in Critical COVID-19: A Retrospective Cohort Study. J Inflamm Res. 2025 Aug 14;18:11139-11153. doi: 10.2147/JIR.S531962. eCollection 2025. PMID 40831520